CLINICAL TRIAL: NCT06720922
Title: Magnetic Resonance-guided Laser Interstitial Thermal Therapy for Mesial Temporal Lobe Epilepsy: A Prospective, Randomized, Open Blinded, End-point Trial
Brief Title: MRgLITT for mTLE: A PROBE Trial
Acronym: MINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Kai Zhang, Dr., Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-073-02
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Temporal Lobe Epilepsy (TLE)
Keywords: Magnetic Resonance-guided Laser Interstitial Thermal Therapy; Open Surgery; Temporal Lobe Epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe | interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Surgery (anterior temporal lobectomy, ATL) (Experimental)
  Interventions: Procedure: Open Surgery
- Minimally Invasive Surgery (MRgLITT) (Active Comparator)
  Interventions: Procedure: Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT)

INTERVENTIONS:
Procedure: Resonance-guided Laser Interstitial Thermal Therapy (MRgLITT) — MRgLITT employs laser energy delivered through a stereotactically placed laser applicator to precisely ablate the epileptogenic tissue.
  Arms: Minimally Invasive Surgery (MRgLITT)
Procedure: Open Surgery — Traditional Open Surgery
  Arms: Open Surgery (anterior temporal lobectomy, ATL)

SUMMARY:
How does magnetic resonance-guided laser interstitial thermal therapy (MRgLITT) impact clinical prognosis in mesial temporal lobe epilepsy (mTLE)?

DETAILED DESCRIPTION:
1. Compare the clinical prognosis between magnetic resonance-guided laser interstitial thermal therapy (MRgLITT) and traditional open surgery (OS) on patients with mesial temporal lobe epilepsy (mTLE).
2. Explore the factors associated with seizure outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years.
* Drug-resistant mesial temporal lobe epilepsy.
* Seizure frequency ≥ 1 time /month.
* Participants approved.

Exclusion Criteria:

* History of brain surgery.
* Intracranial space occupying lesions.
* Individuals with significant medical comorbidities or conditions that pose an excessive risk for surgery, such as severe cardiovascular disease, respiratory disorders, or uncontrolled systemic infections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Seizure freedom rate | 6-month, 1-year after surgery
  According to International League Against Epilepsy [ILAE] Outcome Scale

SECONDARY OUTCOMES:
Seizure frequency | 6-month, 1-year after surgery
  Times/Months
Seizure severity | 6-month, 1-year after surgery
  National Hospital Seizure Severity Scale (NHS3)
Cognitive function evaluation | 6-month, 1-year after surgery
  Multiple Ability Self-Report Questionnaire (MASQ)
Memory function evaluation | 6-month, 1-year after surgery
  Multifactorial Memory Questionnaire (MMQ)
Quality of life for epilepsy patients | 6-month, 1-year after surgery
  EQ-5D-5L
Adverse events | within 7 days, 6-month, 1-year after surgery
  percentage
Severe adverse events | within 7 days, 6-month, 1-year after surgery
  percentage
Length of hospital stay | after surgery
  days
Rate of antiepileptic drug reduction or withdrawn | 1-year after surgery
  percentage
Rate of reoperations | 1-year after surgery
  percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mo J, Guo Z, Wang X, Zhang J, Hu W, Shao X, Sang L, Zheng Z, Zhang C, Zhang K. Magnetic resonance-guided laser interstitial thermal therapy vs. open surgery for drug-resistant mesial temporal lobe epilepsy: a propensity score matched retrospective cohort study. Int J Surg. 2024 Jan 1;110(1):306-314. doi: 10.1097/JS9.0000000000000811. PMID 37800596